CLINICAL TRIAL: NCT00410553
Title: A Phase I Study of Halichondrin B Analog E7389 in Combination With Gemcitabine in Patients With Refractory or Advanced Solid Tumors
Brief Title: Eribulin Mesylate and Gemcitabine Hydrochloride in Treating Patients With Metastatic Solid Tumors or Solid Tumors That Cannot be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00172; NCI-2009-00172 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000520315; PMH-PHL-048; PHL-048 (Other: University Health Network-Princess Margaret Hospital); 7444 (Other: CTEP); N01CM00032 (NIH); N01CM17107 (NIH)
Record Dates: First submitted 2006-12-11; First posted 2006-12-13 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Adult Solid Neoplasm; Recurrent Ovarian Carcinoma; Recurrent Uterine Corpus Carcinoma; Stage III Ovarian Cancer AJCC v6 and v7; Stage III Uterine Corpus Cancer AJCC v7; Stage IV Ovarian Cancer AJCC v6 and v7; Stage IV Uterine Corpus Cancer AJCC v7
MeSH Terms: conditions — Ovarian Neoplasms | interventions — eribulin; Gemcitabine

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): Patients receive eribulin mesylate IV and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 OR on days 1 and 8. Courses repeat every 28 or 21 days* in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Eribulin Mesylate; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Eribulin Mesylate — Given IV
  Other Names: B1939 Mesylate; E7389; ER-086526; Halaven; Halichondrin B Analog
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemzar; LY-188011; LY188011

SUMMARY:
This phase I trial is studying the side effects and best dose of eribulin mesylate and gemcitabine hydrochloride in treating patients with metastatic or unresectable solid tumors. Drugs used in chemotherapy, such as eribulin mesylate and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the recommended phase II dose (RPTD) of E7389 (eribulin mesylate) when given in combination with gemcitabine (gemcitabine hydrochloride) in patients with advanced cancer.

II. Determine the safety, tolerability, and toxicity profile of E7389 and gemcitabine given in combination.

III. Assess the antitumor activity of E7389 in combination with gemcitabine in patients with measurable disease.

IV. Determine the pharmacokinetic profile of E7389 and gemcitabine to assess for any possible interactions between the two agents.

OUTLINE: This is a multicenter, dose-escalation study. Patients receive eribulin mesylate intravenously (IV) and gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 OR on days 1 and 8.

Courses repeat every 28 or 21 days* in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of eribulin mesylate and gemcitabine hydrochloride until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity (DLT). NOTE: *If DLT is observed at the first dose level of the 28-day schedule, subsequent patients are treated on days 1 and 8 of the 21-day schedule; patients enrolled in the expansion cohort (patients with ovarian or endometrial cancer or chemotherapy-naive or minimally pre-treated cancer) receive treatment according to the 21-day schedule.

After completion of study treatment, patients are followed at 4 weeks and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative antineoplastic drug treatments do not exist or are no longer effective:

  * Ovarian/Endometrial Expansion Cohort: Patients must have histologically or cytologically confirmed ovarian or endometrial malignancy that is metastatic or unresectable and for which standard curative antineoplastic drug treatments do not exist or are no longer effective
* CHEMOTHERAPY: Patients may have had up to two prior chemotherapy regimens for advanced or metastatic incurable solid tumors; prior (neo) adjuvant chemotherapy is allowed and not considered among the maximum of two prior regimens; patients must have completed any prior chemotherapy at least 4 weeks prior to registration; prior treatment with gemcitabine is not allowed

  * Chemo Naïve/Minimally Pre-Treated Cohort: Patients may not have received any prior chemotherapy for metastatic disease; prior adjuvant chemotherapy is allowed; patients must have completed any prior chemotherapy at least 4 weeks prior to registration; prior treatment with gemcitabine is not allowed
  * RADIATION: patients may have received prior radiation, however this must have been completed at least 4 weeks prior to registration; patients must not have had more than 40% of their bone marrow irradiated and must have either measurable disease outside the field or progression post radiation therapy
  * SURGERY: patients may have had prior surgery; patients must be at least 4 weeks from any major surgery prior to registration on the study
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2 (Karnofsky >= 60%)
* Life expectancy > 3 months
* Leukocytes >= 3 x 10^9/L
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Since cytochrome P450 (CYP)3A4 appears to be the major enzyme responsible for the human hepatic metabolism of E7389 in vitro, the concurrent use of inhibitors and inducers of CYP3A4 are prohibited during the study treatment period; concurrent use of CYP3A4 substrates are allowed, however, use caution and monitor the patient for potential drug interactions
* The effects of E7389 on the developing human fetus are unknown; for this reason and because antitubulin agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, biologic therapy, hormonal therapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered to < Common Terminology Criteria for Adverse Events (CTCAE) grade 2 from adverse events due to agents administered more than 4 weeks earlier are not eligible to participate in this study; grade 1 persisting toxicities or those deemed irreversible will not be exclusionary; patients who have received prior gemcitabine are also excluded
* Patients may not be receiving any other investigational agents concurrently; patients should not be receiving any other anticancer therapy while on study, such as hormonal, biologic, or targeted therapies
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to E7389 or gemcitabine used in study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because E7389 is an antitubulin agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with E7389, breastfeeding should be discontinued if the mother is treated with E7389; these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with E7389; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-11-14 (Actual); Primary Completion 2012-10-24 (Actual); Study Completion 2012-10-24 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of eribulin mesylate administered with gemcitabine hydrochloride in advanced/metastatic solid tumors | Course 1
  The Common Terminology Criteria for Adverse Events (CTCAE version 3 will be used to grade toxicity.
Recommended phase II dose of eribulin mesylate in combination with gemcitabine hydrochloride | Course 1
  Defined as one dose level below the dose at which 2 or more patients experience a DLT. If =< 1 DLT is observed at dose level 5, then this will be the RPTD.
Safety, tolerability, toxicity profile, and dose-limiting toxicity of eribulin mesylate | From the time of their first treatment with eribulin mesylate
  Graded using the CTCAE version 3.
Pharmacokinetic profiles of eribulin mesylate and gemcitabine hydrochloride | Days 1, 2, 3, 5, and 8 of course 1
  Plasma samples for the determination of eribulin mesylate plasma concentration will be analyzed in conjunction with Eisai Pharmaceuticals. Plasma samples for the determination of gemcitabine plasma concentration will be analyzed through methods developed at the Princess Margaret Hospital.

SECONDARY OUTCOMES:
Preliminary clinical antitumor activity of eribulin mesylate | Baseline, every 2 courses, and 4 weeks post-treatment
  Assessed using radiologic images (CT scans). Measured by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
Objective response rate in patients with measurable disease | Baseline, every 2 courses, and 4 weeks post-treatment
  Measured by RECIST criteria. All tests will be two-sided and a p-value of 0.05 or less will be considered statistically significant. Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest. 95% confidence intervals will be provided for estimates of interest where possible.
Duration of response in patients with measurable disease | From the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented
  Estimated using the Kaplan-Meier method.
Time to disease progression in patients with measurable disease | From start of treatment until the criteria for progression are met
  Estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Rakesh Goel, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (2):
- Canada (2):
  - Ottawa Hospital-Civic Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Lheureux S, Oza AM, Laurie SA, Halford R, Jonker D, Chen E, Keller D, Bourade V, Wang L, Doyle L, Siu LL, Goel R. A phase I combination dose-escalation study of eribulin mesylate and gemcitabine in patients with advanced solid tumours: a study of the Princess Margaret Consortium. Br J Cancer. 2015 Dec 1;113(11):1534-40. doi: 10.1038/bjc.2015.343. Epub 2015 Nov 10. PMID 26554651